CLINICAL TRIAL: NCT07096908
Title: Treatment With Tirzepatide of the Disease of Obesity in People With Type 1 Diabetes
Brief Title: Tirzepatide Use in People With Obesity and Type 1 Diabetes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief of Medical Sector (CMO), Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA HM-2025-03
Record Dates: First submitted 2025-06-25; First posted 2025-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Type1diabetes; Obesity
Keywords: T1D; tirzepatide; weight loss; obesity
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Tirzepatide; Saline Solution

STUDY DESIGN:
Intervention Model Description: The trial is a 76-week, randomized, double-blind, parallel-group, 2- arm, trial comparing maximal tolerable dose of tirzepatide up to 15mg once weekly with placebo once weekly in participants with a BMI ≥27 kg/m2 and T1DM.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide (Experimental): Tirzepatide subcutaneous injections will be given weekly for 76 weeks. Starting dose will be 2.5mg and dose will be increased gradually, by increments of 2.5mg, every 4 weeks to reach 15 mg at week 24 based on patient's tolerability of side effects (i.e. starting dose 2.5 mg, then dose will be increased to 5 mg, 7.5mg,10 mg, 12.5mg then finally 15 mg).
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): an equivalent volume of normal saline 0.9% will be given to the placebo arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — weekly injections
  Arms: Tirzepatide
Drug: Placebo — weekly injections
  Other Names: Normal Saline 0.9%
  Arms: Placebo

SUMMARY:
Tirzepatide, a gut hormone-based medication, has shown promising results in treating obesity, with ~22% weight loss and mild side effects. However, patients with type 2 diabetes typically experience only about 15% weight loss with tirzepatide, despite tolerating the medication well. Its effects in people with both obesity and type 1 diabetes remain largely unknown.

Although tirzepatide is not approved for glycemic control in type 1 diabetes, it is licensed for obesity treatment in Gulf and Europe. In Kuwait, more than a quarter of people with type 1 diabetes also have obesity, presenting a unique opportunity to study tirzepatide's impact.

This randomized, double-blind controlled trial will evaluate the safety and efficacy of tirzepatide in patients with type 1 diabetes and obesity, comparing usual care with the maximum tolerable dose of tirzepatide to assess its impact on weight loss. The findings may help address important safety concerns and have the potential to inform and influence future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities.
2. Male or female, adults.
3. Documented diagnosis of T1DM (per ADA 2024definition/criteria) for at least 1 year before screening visit with C-peptide level of less than 0.01nm/L.
4. Body mass index (BMI) ≥ 27.0 kg/m2
5. History of at least one self-reported unsuccessful dietary effort to lose body weight.
6. Must be using a Continuous Glucose Monitoring (CGM) device for at least 2 months before the screening visit and be willing to wear a CGM device for the duration of the study.

Exclusion Criteria:

1. Diabetes related:

   * Glycated hemoglobin (HbA1c) ≥86 mmol/mol (10%) as measured by the central laboratory at screening.
   * Treatment with a glucagon-like peptide-1 receptor agonist within 180 days before screening.
   * Preproliferative or proliferative retinopathy
   * Experienced diabetic ketoacidosis within 6 months of screening visit.
   * Experienced severe hypoglycemia (Level 3) within 6 months of screening visit.
2. Obesity-related:

   * A self-reported change in body weight >5 kg (11 lbs) within 90 days before screening irrespective of medical records.
   * Treatment with any medication for the indication of obesity within the past 90 days before screening.
   * Previous or planned (during the trial period) obesity treatment with surgery or a weight-loss device. However, the following are allowed: (1) liposuction and/or abdominoplasty, if performed >1 year before screening; (2) lap banding, if the band has been removed >1 year before screening; (3) intragastric balloon, if the balloon has been removed >1 year before screening; or (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed >1 year before screening.
   * Uncontrolled thyroid disease, defined as thyroid stimulating hormone >6.0 mIU/L or <0.4 mIU/L as measured by the central laboratory at screening.
3. Mental health:

   * History of major depressive disorder within 2 years before screening.
   * Diagnosis of other severe psychiatric disorder (e.g. schizophrenia, bipolar disorder).
   * A Patient Health Questionnaire-9 score of ≥15 at screening.
   * A lifetime history of a suicidal attempt.
   * Suicidal behavior within 30 days before screening.
   * Suicidal ideation corresponding to type 4 or 5 on the Columbia-Suicide Severity Rating Scale within the past 30 days before screening.
4. General safety:

   * Use of non-herbal Chinese medicine or other non-herbal local medicine with unknown/unspecified content within 90 days before screening.
   * Presence of acute pancreatitis within the past 180 days prior to the day of screening.
   * History or presence of chronic pancreatitis.
   * Calcitonin ≥100 ng/L as measured by the central laboratory at screening.
   * Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
   * Renal impairment measured as estimated glomerular filtration rate value of <15 mL/min/1.73m2 as defined by KDIGO 2012 by the central laboratory at screening.
   * History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed.
   * Any of the following: myocardial infarction, stroke, hospitalization for unstable angina, or transient ischemic attack within the past 60 days prior to screening.
   * Subject presently classified as being in New York Heart Association Class IV.
   * Surgery scheduled for the duration of the trial, except for minor surgical procedures, in the opinion of the investigator.
   * Known or suspected abuse of alcohol or recreational drugs.
   * Known or suspected hypersensitivity to trial product(s) or related products.
   * Previous participation in this trial. Participation is defined as signed informed consent.
   * Participation in another clinical trial within 90 days before screening.
   * Other subject(s) from the same household participating in any semaglutide trial.
   * Female who is pregnant, breast-feeding, or intends to become pregnant, or is of child-bearing potential and not using a highly effective contraceptive method.
   * Any disorder, unwillingness, or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2028-02-25 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Bodyweight | 76 weeks
  Percent body weight change (%)

SECONDARY OUTCOMES:
HbA1c | 76 weeks
  Change in HbA1c levels (%)
Time in range | 76 weeks
  Change in continuous glucose monitoring (CGM) metrics (time in range (3.9-10mmol/L))
Systolic Blood pressure | 76 weeks
  Change in blood pressure
Diastolic Blood pressure | 76 weeks
  Change in blood pressure
Time in hypoglycaemia | 76 weeks
  Change in continuous glucose monitoring (CGM) metrics (time in hypoglycaemia (mild < 3.9, severe < 2.5mmol/L))
Total cholesterol | 76 weeks
  Change in lipid parameters (total cholesterol)
HDL | 76 weeks
  Change in lipid parameters (HDL)
Triglycerides | 76 weeks
  Change in lipid parameters (Triglycerides)
LDL | 76 weeks
  Change in lipid parameters (LDL)
SF-36 (36-Item Short Form Survey) for Quality of life | 76 weeks
  Quality of life will be assessed using SF-36 questionnaires. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
CRP | 76 week
  Inflammatory markers will be assessed through blood tests.

OTHER OUTCOMES:
Diastolic cardiac function on MRI | 76 weeks
  Diastolic cardiac function on MRI is primarily assessed by analyzing the left ventricular (LV) filling patterns and myocardial mechanics during diastole, the heart's relaxation and filling phase. Left ventricle filling curves will be measured by tracing the endocardial and epicardial borders, Left ventricle volume curves will show the changes in left ventricle volume during diastole.
Liver stiffness | 76 weeks
  Liver stiffness as caused by liver fat will be assessed using MRI
Kidney Disease: Improving Global Outcomes (KDIGO) score for Diabetic nephropathy | 76 weeks
  The KDIGO (Kidney Disease: Improving Global Outcomes) score for diabetic nephropathy will be used as it combines eGFR and urine albumin creatinine ratio. The stages of diabetic nepropathy starts from 1 and increases to 5. A higher score indicates worse diabetic nephropathy.
Diabetic Retinopathy Severity Scale (DRSS) | 76 weeks
  The Diabetic Retinopathy Severity Scale (DRSS) is the primary score used to assess the severity of diabetic retinopathy, according to Retina Today. It ranges from level 10 (normal) to level 85 (advanced proliferative diabetic retinopathy).
Fat mass: fat free mass ratio | 76 weeks
  Body composition will be assessed using dual-energy X-ray absorptiometry (DXA).
Incidence of treatment emergent events | 76 weeks
  Side effects of medications
Functional improvements in quality of life | 76 weeks
  Quality of life will be assessed using SF-36 questionnaires. Scores for the functional domain range from 0 to 100, with a higher score defining a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa Al Ozairi, MD, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Sharq, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided